CLINICAL TRIAL: NCT00774423
Title: Multicentric, Randomized, Double-blind Study Versus Placebo, With Two Parallel Groups Treated to Evaluate the Efficacy and the Tolerance of Riluzole in Children and Young Adults (6 to 20 Years of Age) With SMA. (Type II and Type III)
Brief Title: Study to Evaluate the Efficacy of Riluzole in Children and Young Adults With Spinal Muscular Atrophy (SMA)
Acronym: ASIRI
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P040904
Record Dates: First submitted 2008-10-16; First posted 2008-10-17 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2011-09

CONDITIONS: SMA
Keywords: Spinal muscular atrophies (SMA); Degeneration of the motor neurons; Anterior horn of the spinal cord; Riluzole
MeSH Terms: interventions — Riluzole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): MAIN EXCIPIENT OF THE RILUTEK
  Interventions: Drug: Riluzole
- Riluzole (Active Comparator): RILUTEK
  Interventions: Drug: Riluzole

INTERVENTIONS:
Drug: Riluzole — 50 mg per day during 24 months

SUMMARY:
This is a multicentric, randomized, double-blind study versus placebo, with two parallel groups treated to evaluate the efficacy and the tolerance of Riluzole in children and young adults (6 to 20 years of age) with SMA. (Type II and Type III).

DETAILED DESCRIPTION:
ASIRI study should allow to evaluate the efficacy and the tolerance of Riluzole in children and young adults (6 to 20 years of age) with SMA. This is a multicentric, randomized, double-blind study versus placebo, with two parallel groups treated and followed during 2 years. It has been preceded by a 7 days pharmacokinetic phase, concerning 14 patients, aiming to provide information on the kinetic profile of Riluzole in children. The drug could stabilize patients condition, and especially interrupt paralysis progression; those are the desired effects.

There is an open-label study of the long term safety of riluzole therapy in spinal muscular atrophies types II and III, with patients previously enrolled in ASIRI double-blind study.

ELIGIBILITY:
Inclusion Criteria:

* Patients afflicted with spinal muscular atrophy, type II or III, with genetic defect confirmed.
* Age between 6 and 20 years old.
* Score MFM at least 12
* Negative pregnancy test for women of child-bearing age
* Signing of an informed consent form, after appropriate information has been provided (if the patient is under 18 years old, both parents are required to sign the form too; otherwise, only her (his) agreement is necessary).

Exclusion Criteria:

* Patients already treated with Riluzole
* Concomitant treatment with: GAPAPENTINE, DEXTROMETHORPHANE, amantadine, any hepatotoxic medication that cannot be stopped, any other experimental product
* Hepatic insufficiency: SGPT and/or SGOT levels higher than or equal to twice the normal higher limit
* Renal insufficiency (creatinine above 115 micromoles/l)
* Severe cardiac insufficiency
* Current pneumopathy (clinical signs of an acute episode, confirmed by pulmonary X-ray, requiring specific treatment)
* Pregnancy or nursing for women; non-abstinence or absence of effective contraception for nubile women
* Any pathology or other circumstance likely to interfere with a regular follow-up
* No affiliation to any social insurance system

Ages: 6 Years to 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 141 (Actual)
Dates: Start 2006-01; Primary Completion 2011-09 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
The drug could stabilize patients condition during 24 months, and especially interrupt paralysis progression: Motor function (MFM scale) | 6, 12, 18 and 24 months

SECONDARY OUTCOMES:
Forced vital capacity (spirometry) | 6, 12, 18 and 24 months
Quality of life (OKado questionnaire) | 12 and 24 months
Measure of functional independence (MFI) | 6,12,18 and 24 months
Tolerance evaluation: Somatic symptoms and adverse events Blood pressure and heart rate Weight and size Blood count, hepatic enzymes and bilirubin | every 3 months

CONTACTS AND LOCATIONS:
Overall Officials: BRIGITTE ESTOURNET, PU-PH, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- Hopital Raymond Poincare, Garches, France